CLINICAL TRIAL: NCT03467815
Title: Wireless Assessment of Respiratory and Circulatory Distress in Chronic Obstructive Pulmonary Disease - A Pilot Study
Brief Title: Wireless Assessment of Respiratory and Circulatory Distress in Chronic Obstructive Pulmonary Disease
Acronym: WARD-COPD
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Technical University of Denmark (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mikkel Elvekjaer, M.D., Bispebjerg Hospital
Other Study IDs: Bispebjerg Hospital Research
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Dyspnea
Keywords: Wireless monitoring; Continuous monitoring; Vital parameters; Clinical deterioration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For patients admitted to the medical ward, it is usually difficult to predict if their clinical condition will deteriorate, however subtle changes in vital signs are usually present 8 to 24 hours before a life-threatening event such as respiratory failure leading to ICU admission, or unanticipated cardiac arrest. Such adverse trends in clinical observations can be missed, misinterpreted or not appreciated as urgent. New continuous and wearable 24/7 clinical vital parameter monitoring systems offer a unique possibility to identify clinical deterioration before patients progress beyond the point-of-no-return, where adverse events are inevitable. The WARD-COPD project aims to determine the number and duration of cardiopulmonary micro events during the first 4 days after hospital admission with Acute Exacerbation of COPD. We will also test the server installation, develop a database of core data and assess the frequency of artefacts and failure to capture the continuous monitoring signal.

ELIGIBILITY:
Inclusion Criteria:

Adult patients admitted to hospital for Acute Exacerbation of COPD (AECOPD). Investigators will review the electronic patient chart for a primary diagnosis of AECOPD.

Exclusion Criteria:

* Patient expected not to cooperate.
* Patient allergic to plaster, plastic or silicone.
* Active therapy withdrawn

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to hospital for Acute Exacerbation of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Blood oxygen saturation resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  Hypoxemia: arterial oxygen saturation < 92 %
Heart rate resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  All data from the monitoring will be analyzed using the thresholds from the EWS algorithm and will be sorted into relevant categories. The following thresholds are used:
  Bradycardia: pulse < 41 bpm Tachycardia: pulse > 130 bpm
Respiratory rate resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  Bradypnea: < 9 breaths/min Tachypnea: > 24 breaths/min
Blood pressure resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  Hypotension: Systolic blood pressure < 91 mmHg Hypertension: Systolic blood pressure > 219 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark